CLINICAL TRIAL: NCT03223701
Title: Efficacy Study Using Solum IV, Bone Marrow Concentrate With General Fluid Concentrate in Transforaminal Lumbar Interbody Fusion
Brief Title: Efficacy of Using Solum IV and BMC With GFC in TLIF
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was never initiated due to contracting issues
Sponsor: Seton Healthcare Family (Other)
Collaborators: Celling Biosciences (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-17-101
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Degenerative Disc Disease; Isthmic-lytic Spondylolisthesis; Degenerative Spondylolisthesis; Spinal Stenosis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center clinical study. Ten patients will be enrolled and undergo an Transforaminal Lumbar Interbody Fusion (TLIF) with a spinal fixation system and receive Solum IV (Celling Biosciences) and patient's bone marrow concentrate with general fluid concentrate (GFC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment group (Other): The group will consist of 10 patients who would be examined for fusion rates of Transforaminal Lumbar Interbody Fusion with a standalone lumbar implant device and Solum IV and the patient's bone marrow concentrate and general fluid concentrate.
  Interventions: Combination Product: Solum IV, Bone Marrow Concentrate with general fluid concentrate (GFC) in Transforaminal Lumbar Interbody Fusion

INTERVENTIONS:
Combination Product: Solum IV, Bone Marrow Concentrate with general fluid concentrate (GFC) in Transforaminal Lumbar Interbody Fusion — The bone marrow aspirate (BMA) will be taken from the iliac crest of the enrolled subjects. The BMA will be transferred to a processor that will use ART BMC Plus (Celling Biosciences, Austin, TX) platform technology to obtain the BMC preparation. The plasma component that remains as a by-product of generating the BMC will then be concentrated by the ART BMC Plus device to create a concentrated plasma/general fluid concentrate (GFC). The enrolled subjects' BMC and GFC will be provided to the principle investigator who will combine the two together with Solum IV using the Graft Delivery Kit (Celling Biosciences) and perform a TLIF procedure. (See Appendix B for Graft Delivery Kit). All subjects will be assigned to receive lumbar interbody fusion via a TLIF approach with Solum IV bone graft and BMC with GFC in the interbody space of a TLIF using cynch bullet cage (@SpineSmith) and Stryker based pedicle screw system (Xia 3 system).

SUMMARY:
The purpose of this study is to examine the efficacy of using Solum IV and bone marrow concentrate with general fluid concentrate in Transforaminal Lumbar Interbody Fusion (TLIF).

DETAILED DESCRIPTION:
This is a prospective, single-center clinical study. Ten patients will be enrolled and undergo an TLIF with a spinal fixation system and receive Solum IV (Celling Biosciences) and patient's BMC with GFC.

The bone marrow aspirate (BMA) will be taken from the iliac crest of the enrolled subjects. The BMA will be transferred to a processor that will use ART BMC Plus (Celling Biosciences, Austin, TX) platform technology to obtain the BMC preparation. The plasma component that remains as a by-product of generating the BMC will then be concentrated by the ART BMC Plus device to create a concentrated plasma/general fluid concentrate (GFC). The enrolled subjects' BMC and GFC will be provided to the principle investigator who will combine the two together with Solum IV using the Graft Delivery Kit (Celling Biosciences) and perform a TLIF procedure. (See Appendix B for Graft Delivery Kit). All subjects will be assigned to receive lumbar interbody fusion via a TLIF approach with Solum IV bone graft and BMC with GFC in the interbody space of a TLIF using cynch bullet cage (@SpineSmith) and Stryker based pedicle screw system (Xia 3 system).

All study subjects will be assessed for fusion rate, complication rates and subject-reported outcomes at designated intervals up to 12 months after surgery. X-rays (anterior-posterior, lateral, flexion-extension) will be taken at pre-operatively, 3, 6, and 12 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is skeletally mature and older than 18 years of age
2. One and contiguous 2 or 3 level primary lumbar fusions.
3. L1 to S1 with a primary diagnosis of one or more of the following:

   1. Degenerative disc disease,
   2. Isthmic-lytic spondylolisthesis,
   3. Degenerative spondylolisthesis
   4. Spinal stenosis.
4. Subject has received conservative (non -surgical treatment for back pain for a minimum of 6 months and is unresponsive
5. Subject understand the conditions of enrollment and is willing to sign and date the informed consent form
6. Subject agrees to comply with study visits

   -

Exclusion Criteria:

1. Previous bilateral Iliac Crest Bone Graft (ICBG) harvest
2. Previous instrumented fusion at the same or adjacent level
3. Active systemic infection, infection localized to the site of implantation or at aspiration site
4. Vulnerable patients

   1. Nursing home residents
   2. Prisoners
   3. Other institutionalized persons
   4. Persons with decisional incapacity
5. Pregnant women or interested in becoming pregnant in the next 12 months
6. Subjects with certain autoimmune diseases (such as lupus)
7. Subject has progressive neuromuscular disease
8. Active hepatitis, AIDS, ARS or is HIV positive
9. Syringomyelia at any spinal levels
10. Any other condition that would interfere with the subject self-assessment of pain, function or quality of life
11. Subjects with multiple allergies
12. Subjects with any history of cancer (except for basal cell carcinoma of the skin)
13. Significant osteoporosis
14. Subject is younger than or equal to 18 years of age
15. Subjects with a BMI of 40 or greater
16. Subject has diabetes mellitus requiring daily insulin management
17. Subject has allergy to implant materials (such as titanium, titanium alloy)
18. Subject has primary or metastatic tumors involving the spine
19. Subject is participating in another investigational study for a similar purpose
20. Subject has a history of significant mental illness or mental incapacity
21. Subject is currently smoker and will not cease smoking from the time of study enrollment up through 3 months post-operatively, nicotine users for whom post-operative bone stimulation would be prescribed, or has a recent history of alcohol or other substance abuse within the past 2 years
22. Subject is receiving workers compensation
23. Absence of English language reading or writing skills

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-30 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Radiological assessment : Fusion Status | 3 months post-treatment
  X-rays (anterior-posterior, lateral, flexion-extension)
Radiological assessment : Fusion Status | 6 months post-treatment
  X-rays (anterior-posterior, lateral, flexion-extension)
Radiological assessment : Fusion Status | 12 months post-treatment
  X-rays (anterior-posterior, lateral, flexion-extension)

SECONDARY OUTCOMES:
Visual Analog Scale | Pre-treatment
  Patient reported pain score
Visual Analog Scale | 3 months post-treatment
  Patient reported pain score
Visual Analog Scale | 6 months post-treatment
  Patient reported pain score
Visual Analog Scale | 12 months post-treatment
  Patient reported pain score
Oswestry Disability Index | Pre-treatment
  Patient reported disability score
Oswestry Disability Index | 3 months post-treatment
  Patient reported disability score
Oswestry Disability Index | 6 months post-treatment
  Patient reported disability score
Oswestry Disability Index | 12 months post-treatment
  Patient reported disability score

CONTACTS AND LOCATIONS:
Overall Officials: Eeric Truumees, MD, Principal Investigator — Seton Spine and Scoliosis Center
Locations (1):
- Seton Spine and Scoliosis Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hernigou P, Beaujean F. Treatment of osteonecrosis with autologous bone marrow grafting. Clin Orthop Relat Res. 2002 Dec;(405):14-23. doi: 10.1097/00003086-200212000-00003. PMID 12461352
- [Background] Gan Y, Dai K, Zhang P, Tang T, Zhu Z, Lu J. The clinical use of enriched bone marrow stem cells combined with porous beta-tricalcium phosphate in posterior spinal fusion. Biomaterials. 2008 Oct;29(29):3973-82. doi: 10.1016/j.biomaterials.2008.06.026. Epub 2008 Jul 18. PMID 18639333
- [Background] Galois L, Bensoussan D, Diligent J, Pinzano A, Henrionnet C, Choufani E, Stoltz JF, Mainard D. Autologous bone marrow graft and treatment of delayed and non-unions of long bones: technical aspects. Biomed Mater Eng. 2009;19(4-5):277-81. doi: 10.3233/BME-2009-0592. PMID 20042794
- [Background] Johnson RG. Bone marrow concentrate with allograft equivalent to autograft in lumbar fusions. Spine (Phila Pa 1976). 2014 Apr 20;39(9):695-700. doi: 10.1097/BRS.0000000000000254. PMID 24503679
- [Result] Hernigou P, Poignard A, Beaujean F, Rouard H. Percutaneous autologous bone-marrow grafting for nonunions. Influence of the number and concentration of progenitor cells. J Bone Joint Surg Am. 2005 Jul;87(7):1430-7. doi: 10.2106/JBJS.D.02215. PMID 15995108